CLINICAL TRIAL: NCT05954689
Title: Femoral Artery Block for Reduction of Tourniquet Induced Hypertension: a Randomised Controlled Trial
Brief Title: Femoral Artery Block for Reduction of Tourniquet Induced Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital da Luz, Portugal (Other)
Responsible Party: Principal Investigator, Vasyl Katerenchuk, Anaesthesiology Resident, Hospital da Luz, Portugal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U1111-1293-7325
Record Dates: First submitted 2023-07-06; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Tourniquets; Anesthesia, Conduction; Anesthetics, Local; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral artery block (Experimental): An experienced Anesthesiologist will perform the femoral blocks, under ultrasound guidance with a linear probe and a 50mm (millimeters) or 80mm needle. No nerve stimulator will be used during the block. In both groups, femoral nerve block at the nerve sheath will be performed with 20mL (milliliters) 0.5% ropivacaine. In the interventional group, additionally to the previous block, the needle will be retracted and advanced to the antero-medial side of the femoral artery where 10mL 0.5% ropivacaine will be injected after negative aspiration.
  Interventions: Other: Femoral artery block
- No intervention (No Intervention)

INTERVENTIONS:
Other: Femoral artery block — Injection on the antero-medial side of the femoral artery of 10mL 0.5% ropivacaine with ultrasound guidance.
  Arms: Femoral artery block

SUMMARY:
A randomised controlled trial to assess the impact of femoral artery block on the incidence of tourniquet hypertension in patients receiving cruciate ligament surgery with > 30 minutes of tourniquet under combined anaesthesia (balanced general anaesthesia and femoral nerve blocks).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I to III
* Receiving cruciate ligament surgery with > 30 minutes of tourniquet
* Combined anesthesia (balanced general anesthesia and femoral nerve block)

Exclusion Criteria:

* Nerve block contraindications (block site infection, allergic to local anesthetic)
* Tourniquet contraindications (peripheral vascular disease or neuropathy, previous arterial bypass graft)
* Tourniquet inflation time < 30 min
* Patient refusal
* Pregnant patients
* Patients with a active psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-10 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Tourniquet Hypertension (TH) | Thought intra-operative time (after induction of anesthesia and until emergence from anesthesia)
  Defined as Systolic Blood Pressure (SBP) increased >30% after 30 minutes of tourniquet
Systolic blood pressure 30 minutes after tourniquet inflation | 30 minutes after tourniquet inflation
  SBP at 30 minutes after tourniquet inflation
Systolic blood pressure 45 minutes after tourniquet inflation | 45 minutes after tourniquet inflation
  SBP at 45 minutes after tourniquet inflation
Systolic blood pressure 60 minutes after tourniquet inflation | 60 minutes after tourniquet inflation
  SBP at 60 minutes after tourniquet inflation
Systolic blood pressure 75 minutes after tourniquet inflation | 75 minutes after tourniquet inflation
  SBP at 75 minutes after tourniquet inflation
Systolic blood pressure 90 minutes after tourniquet inflation | 90 minutes after tourniquet inflation
  SBP at 90 minutes after tourniquet inflation
Systolic blood pressure 115 minutes after tourniquet inflation | 115 minutes after tourniquet inflation
  SBP at 115 minutes after tourniquet inflation
Systolic blood pressure 130 minutes after tourniquet inflation | 130 minutes after tourniquet inflation
  SBP at 130 minutes after tourniquet inflation
Mean arterial pressure (MAP) 30 minutes after tourniquet inflation | 30 minutes after tourniquet inflation
  MAP at 30 minutes after tourniquet inflation
Mean arterial pressure 45 minutes after tourniquet inflation | 45 minutes after tourniquet inflation
  MAP at 45 minutes after tourniquet inflation
Mean arterial pressure 60 minutes after tourniquet inflation | 60 minutes after tourniquet inflation
  MAP at 60 minutes after tourniquet inflation
Mean arterial pressure 75 minutes after tourniquet inflation | 75 minutes after tourniquet inflation
  MAP at 75 minutes after tourniquet inflation
Mean arterial pressure 90 minutes after tourniquet inflation | 90 minutes after tourniquet inflation
  MAP at 90 minutes after tourniquet inflation
Mean arterial pressure 115 minutes after tourniquet inflation | 115 minutes after tourniquet inflation
  MAP at 115 minutes after tourniquet inflation
Mean arterial pressure 130 minutes after tourniquet inflation | 130 minutes after tourniquet inflation
  MAP at 130 minutes after tourniquet inflation
Systolic blood pressure variation from baseline at 30 minutes after tourniquet inflation | 30 minutes after tourniquet inflation
  Variation of SBP compared to baseline at 30 minutes after tourniquet inflation
Systolic blood pressure variation from baseline at 45 minutes after tourniquet inflation | 45 minutes after tourniquet inflation
  Variation of SBP compared to baseline at 45 minutes after tourniquet inflation
Systolic blood pressure variation from baseline at 60 minutes after tourniquet inflation | 60 minutes after tourniquet inflation
  Variation of SBP compared to baseline at 60 minutes after tourniquet inflation
Systolic blood pressure variation from baseline at 75 minutes after tourniquet inflation | 75 minutes after tourniquet inflation
  Variation of SBP compared to baseline at 75 minutes after tourniquet inflation
Systolic blood pressure variation from baseline at 90 minutes after tourniquet inflation | 90 minutes after tourniquet inflation
  Variation of SBP compared to baseline at 90 minutes after tourniquet inflation
Systolic blood pressure variation from baseline at 115 minutes after tourniquet inflation | 115 minutes after tourniquet inflation
  Variation of SBP compared to baseline at 115 minutes after tourniquet inflation
Systolic blood pressure variation from baseline at 130 minutes after tourniquet inflation | 130 minutes after tourniquet inflation
  Variation of SBP compared to baseline at 130 minutes after tourniquet inflation
Mean arterial pressure variation from baseline at 30 minutes after tourniquet inflation | 30 minutes after tourniquet inflation
  Variation of MAP compared to baseline at 30 minutes after tourniquet inflation
Mean arterial pressure variation from baseline at 45 minutes after tourniquet inflation | 45 minutes after tourniquet inflation
  Variation of MAP compared to baseline at 45 minutes after tourniquet inflation
Mean arterial pressure variation from baseline at 60 minutes after tourniquet inflation | 60 minutes after tourniquet inflation
  Variation of MAP compared to baseline at 60 minutes after tourniquet inflation
Mean arterial pressure variation from baseline at 75 minutes after tourniquet inflation | 75 minutes after tourniquet inflation
  Variation of MAP compared to baseline at 75 minutes after tourniquet inflation
Mean arterial pressure variation from baseline at 90 minutes after tourniquet inflation | 90 minutes after tourniquet inflation
  Variation of MAP compared to baseline at 90 minutes after tourniquet inflation
Mean arterial pressure variation from baseline at 115 minutes after tourniquet inflation | 115 minutes after tourniquet inflation
  Variation of MAP compared to baseline at 115 minutes after tourniquet inflation
Mean arterial pressure variation from baseline at 130 minutes after tourniquet inflation | 130 minutes after tourniquet inflation
  Variation of MAP compared to baseline at 130 minutes after tourniquet inflation

SECONDARY OUTCOMES:
Isosorbide dinitrate administered for TH | Thought intra-operative time (after induction of anesthesia and until emergence from anesthesia) )
  mg of isosorbide dinitrate administered for TH
Numerical verbal pain scores | Up to 2 hours after emergence from anesthesia
  Numerical verbal pain scores (from 0 to 10, 10 meaning higher pain) assessed 1 hour after emergence of anesthesia in the post-operative care unit (PACU)
Patient post-operative satisfaction | Up to 2 hours after emergence from anesthesia
  Patient post-operative satisfaction with pain treatment measured 1 hour after emergence of anesthesia in the post-operative care unit using a 5-point Likert-scale, namely: 1 - very unsatisfied, 2 - unsatisfied, 3 - neutral, 4 - satisfied, 5 - very satisfied (with higher scores meaning a higher outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Filipa Duarte, Principal Investigator — Hospital da Luz, Lisboa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo YX, Wang GY, Cheng WJ, Yan CZ, Zhao S, Li Z, Liu P, Wang XL. Activation of Opioid Receptors Attenuates Ischemia/Reperfusion Injury in Skeletal Muscle Induced by Tourniquet Placement. Mediators Inflamm. 2021 Jan 15;2021:6699499. doi: 10.1155/2021/6699499. eCollection 2021. PMID 33510583
- [Background] Xu F, Wang X, Li Y, Gao F, Yin C, Yu J, Li W, Zhu L, Wang Q. Combined femoral artery block and femoral nerve block reduces thigh tourniquet-induced hypertension. J Clin Anesth. 2023 May;85:111039. doi: 10.1016/j.jclinane.2022.111039. Epub 2022 Dec 20. PMID 36549034
- [Background] Wahal C, Grant SA, Gadsden J, Rambhia MT, Bullock WM. Femoral artery block (FAB) attenuates thigh tourniquet-induced hypertension: a prospective randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2021 Mar;46(3):228-232. doi: 10.1136/rapm-2020-102113. Epub 2021 Jan 11. PMID 33431616